CLINICAL TRIAL: NCT06133218
Title: Patient-reported Experience and Symptom Measures on Prophylactic Use of Mepitel Film During Post-operative Breast Irradiation - a Danish Intra-patient Randomized Multicentre Study
Brief Title: Patient Reported Outcomes Using Mepitel Film During Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Herning Hospital (Other); Vejle Hospital (Other)
Responsible Party: Principal Investigator, Pia Krause Møller, Clinical Nurse Specialist, MPH, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OP_168
Record Dates: First submitted 2018-03-26; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Radiodermatitis; Breast Neoplasms; Side Effect
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention side - Mepitel Film (Active Comparator): This was an intra-patient randomized study. The patient was randomized for Mepitel film (barrier film) applied on the medial or lateral side of their breast or chest wall during the entire course of radiotherapy; making the patients their own control.
  Interventions: Other: Mepitel Film
- Control side - standard care (No Intervention): The other side of the breast or chest wall is the intra-patient control as the skin on this side was treated according to standard guidelines for skin care during radiotherapy when symptoms or skin reactions occured.

INTERVENTIONS:
Other: Mepitel Film — A safetac-based barrier film with a clinically insignificant bolus effect to protect the skin during radiotherapy.
  Arms: Intervention side - Mepitel Film

SUMMARY:
Breast cancer patients in post-operative radiotherapy (RT) often experience acute skin reactions like erythema, pain, itching and oversensitivity. In 2014 a New Zealand randomized controlled trial (RCT) investigated the prophylactic use of safetac-based film, Mepitel Film, on half of the breast during RT compared to cream, resulting in significant differences in skin moist desquamation (0% vs. 26%). Despite changes in treatment modalities in Denmark toward lower total RT doses, the level of RT-induced skin toxicity could still be of great importance for the patients. The aim of this study is patient-reported symptoms and patient-reported experiences with the prophylactic use of Mepitel Film compared to standard cream treatment.

DETAILED DESCRIPTION:
Aim:

The use of Mepitel Film in the RCT from New Zealand resulted in significant differences in the acute morbidity of the skin. However, the clinical experience in Denmark with the new RT treatment modalities for breast cancer patients with lower total doses and less treatment fractions indicate less severe skin toxicity than the old treatment modalities.

The primary endpoint of this study is to investigate if prophylactic use of Mepitel Film to prevent severe skin reactions makes a difference for the patient experience of their RT induced skin reactions compared to treating the symptoms when they appear according to present clinical guidelines. Additional to the patient-reported experiences with the prophylactic use of Mepitel Film, the patients are asked to report their acute symptoms from the skin in the area with or without Mepitel Film at the end of treatment and two weeks after treatment. A secondary endpoint was a blinded radiotherapy staff evaluation of dermatitis.

Method:

The study was a multicenter trial with participation of three Danish hospitals: Aarhus University Hospital (Herning site), Vejle Hospital, and Odense University Hospital.

For all patients either the lateral or medial part of the treatment area was covered by film based on a randomization; making the patients their own control.

The randomization procedure was conducted by assigned radiotherapists (RTTs) at each hospital in the online system RedCap (Research Electronic Data Capture) provided by Odense Patient Data Explorative Network (OPEN). A block randomization was conducted stratifying for hospital to balance at each institution the number of patients having film applied at the medial or lateral part of the chest.

A questionnaire was developed.consisting of four sections. Two sections with patient-reported outcome measures (PROM) regarding skin symptoms. Furthermore, a section with patient-reported experience measures (PREM) related to the use and preference of the barrier film and finally a section for staff evaluation of dermatitis.

The PROM-questionnaire was developed guided by existing validated questionnaires (RISRAS-scale [14], and the breast cancer specific EORTC-questionnaire [15]). The answers were categorized on a 4-Point Likert Scale (not at all, a little, some, a lot).

The PREM-questionnaire consisted of seven questions regarding comfort and preferences with a 4-point Likert scale (strongly agree, mildly agree, mildly disagree, strongly disagree) and a scale for grading overall health and overall QOL. The questionnaires were cognitively validated by 3 patients.

The patients were asked to fill out the paper-based questionnaire on the day of their final radiotherapy treatment and a similar one at the two week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All women referred to postoperative adjuvant radiotherapy for breast cancer from October 1st 2015 to February 29th 2016 at the three radiotherapy departments.
* Who read and understand Danish
* Patients must have signed and dated a written informed consent form in accordance with regulatory and institutional guidelines.
* Patients must be willing and able to comply the questionnaires and attend a two-week follow-up posttreatment.

Exclusion Criteria:

* Patients included in the ongoing Danish HYPO PBI protocol (hypofractionated partial breast irradiation)

Ages: 18 Years to 125 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Patient-reported experience measures (PREM) | Two-week follow-up after RT
  Patient experiences and preferences regarding Mepitel film for women with breast cancer undergoing radiotherapy based on their own experience with skin toxicity. The PREM-questionnaire consisted of seven questions regarding comfort and preferences with a 4-point Likert scale (strongly agree, mildly agree, mildly disagree, strongly disagree).
Patient-reported outcome measures (PRO) | Two-week follow-up after RT
  The proportion of radiation-induced symptoms with or without film (pain, itching, burning sensation, edema, sensitive or flaky skin) and the effect on work/daily activities measured with a 4-Point Likert Scale (not at all, a little, some, a lot).

SECONDARY OUTCOMES:
Radiodermatitis | Last 1 day of radiotherapy
  The grade of radiodermatitis (RTOG-scale)on the chest side with Mepitel Film vs the skin area treated according to standard care. A blinded evaluation.
Radiodermatitis | Two-week follow-up
  The grade of radiodermatitis (RTOG-scale)on the chest side with Mepitel Film vs the skin area treated according to standard care. A blinded evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Pia K Moeller, MPH, Principal Investigator — Odense University Hospital (OUH)

IPD SHARING:
Plan to Share IPD: No